CLINICAL TRIAL: NCT03107663
Title: A Phase I Study of Positron Emission Tomography (PET/CT) With ⁸⁹Zr-Df-IAB22M2C in Patients With Selected Solid Malignancies (Non Small Cell Lung Cancer (NSCLC), Small Cell Lung Cancer (SCLC), Squamous Cell Carcinoma Head and Neck (SqCCHN), Melanoma, Merkel Cell Tumor, Renal, Bladder, Hepatocellular, Triple Negative Breast, or Gastroesophageal Cancer) or Hodgkin's Lymphoma
Brief Title: ⁸⁹Zr-Df-IAB22M2C PET/CT in Patients With Selected Solid Malignancies or Hodgkin's Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ImaginAb, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2015-22M2C-01.02
Record Dates: First submitted 2017-01-16; First posted 2017-04-11 (Actual); Last update posted 2018-09-18 (Actual); Status verified 2018-09

CONDITIONS: Positron-Emission Tomography; Immunomodulation; Metastatic Solid Malignancies; Hodgkin Lymphoma
Keywords: PET/CT; Imaging; ⁸⁹Zr-Df-IAB22M2C; CD8 + T Cells; Standard of Care
MeSH Terms: conditions — Hodgkin Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ⁸⁹Zr-Df-IAB22M2C Infusion (Experimental): 3.0 (±20%) mCi of ⁸⁹Zr-Df-IAB22M2C (with 0.2 mg, 0.5 mg, 1.0mg, 1.5 mg, 5.0 mg, or 10.0 mg of protein) will be administered intravenously over 5-10 minutes
  Interventions: Drug: ⁸⁹Zr-Df-IAB22M2C Infusion

INTERVENTIONS:
Drug: ⁸⁹Zr-Df-IAB22M2C Infusion — A single dose of 3.0 (±20%) mCi of ⁸⁹Zr-Df-IAB22M2C (with 0.2 mg, 0.5 mg, 1.0mg, 1.5 mg, 5.0 mg, or 10.0 mg of protein) will be administered intravenously over 5-10 minutes.

SUMMARY:
To determine the safety and feasibility of 89Zr-Df-IAB22M2C as an immunoPET tracer; determine the best time window and protein dose for imaging; determine the pharmacokinetic (PK) and biodistribution of the probe; and to determine imaging parameters for optimal lymphoid and tumor visualization.

DETAILED DESCRIPTION:
This is a phase I study of positron emission tomography (PET/CT) with ⁸⁹Zr-Df-IAB22M2C in patients with selected solid malignancies (NSCLC, SCLC, SqCCHN, melanoma, merkel cell tumor, renal, bladder, hepatocellular, triple negative breast, or gastroesophageal cancer) or Hodgkin's lymphoma. Up to 24 subjects are planned to be enrolled in this clinical study.

This phase 1 study is a dose escalation study of ⁸⁹Zr-Df-IAB22M2C to evaluate safety, tolerability, optimal time window and protein dose for imaging, biodistribution, radiation dosimetry, as well as the ability of ⁸⁹Zr-Df-IAB22M2C to detect CD8+ expressing T cells. The investigational imaging agent to be administered in this study will be 3.0 (±20%) mCi dose of ⁸⁹Zr-Df-IAB22M2C injected intravenously. Up to six cohorts of up to 6 patients each will be studied sequentially with dose escalation at 0.2 mg, 0.5 mg, 1.0 mg, 1.5 mg, 5.0 mg, and 10.0 mg total protein doses followed by an optimal dose expansion cohort. Safety as well as lymphoid visualization (LV) on imaging (i.e. signal in tumor and lymphoid organs including spleen, lymph nodes and bone marrow) will be evaluated to drive dose escalation/de-escalation.

At least 2 weeks will separate the ⁸⁹Zr-Df-IAB22M2C administration in the first patient and subsequent patients of each dose cohort to provide an opportunity to detect any acute reaction to the study drug and any adverse events. Tracer administration for subsequent patients in each cohort will be separated by a minimum of 24 hours

Each patient will undergo five (5) post infusion PET/CT scans ( 1 - 2 hours, 6-8 hrs (optional), 24 ± 4 hours, 48 ± 4 hours and 92 - 144 hours).

Pharmacokinetic blood samples will be drawn at the following timepoints: pre-infusion; then post-infusion at 5-10 min, 30 (+/-10) min, 60 (+/- 10) min, 120 (+/- 10) min, 240 (+/- 10) min, 350-490 (+/- 10) min (optional), 24 hrs (visit 3), 48 hrs (visit 4), 92-144 hrs (visit 5). The imaging data collected across the dosing cohort and time series of PET/CT scans will assess biodistribution, dosimetry, and be used to recommend a protein dose and an optimal time window for imaging in future studies

ELIGIBILITY:
Inclusion Criteria:

1. Patients with selected solid malignancies (NSCLC, SCLC, SqCCHN, melanoma, merkel cell tumor, renal, bladder, hepatocellular, triple negative breast, or gastroesophageal cancer) or Hodgkin's lymphoma
2. At least 1 measurable lesion documented on CT/MRI (RECIST criteria 1.1)
3. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2 (Appendix B: ECOG Scoring)
4. Age ≥ 18 years
5. Ability to understand the purposes and risks of the trial and has signed a IRB-approved informed consent form
6. Willingness and ability to comply with all protocol required procedures
7. For men and women of child-bearing potential, use of effective contraceptive methods during the study

Exclusion Criteria:

Patients meeting any of the following criteria will not be eligible for study entry:

1. Known infection with human immunodeficiency virus (HIV)
2. Serious nonmalignant disease or conditions that in the opinion of the investigator and/or ImaginAb could compromise protocol objectives
3. Patients who have had splenectomy.
4. Patients who have any splenic disorders that in the opinion of the investigator and/or ImaginAb could compromise protocol objectives.
5. Patients who are currently receiving any other investigational agent
6. Pregnant women or nursing mothers
7. Hepatic laboratory values:

   1. Bilirubin > 1.5 x ULN (institutional upper limits of normal)
   2. Albumin < 2 g/dL
   3. Other local safety laboratory test results (clinical chemistry and hematology) are determined to be exclusionary by the Investigator.
8. Known sensitivity to glutamic acid or glutamate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-06-19 (Actual); Primary Completion 2018-08-16 (Actual); Study Completion 2018-08-16 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of ⁸⁹Zr-Df-IAB22M2C assessed by local and systemic signs and symptoms of infusion reactions,incidence of adverse events,changes in laboratory test results,dose limiting toxicities,vital signs and 12-lead electrocardiogram findings | From infusion of ⁸⁹Zr-Df-IAB22M2C up to 12 weeks

SECONDARY OUTCOMES:
Evaluate imaging time window with ⁸⁹Zr-Df-IAB22M2C | From infusion of ⁸⁹Zr-Df-IAB22M2C through up to Day 6
Evaluate protein dose for imaging with ⁸⁹Zr-Df-IAB22M2C | From infusion of ⁸⁹Zr-Df-IAB22M2C through up to Day 6
Evaluate the radioactive pharmacokinetics of ⁸⁹Zr-Df-IAB22M2C by determining the time-activity curves for serum (% injected dose/liter), AUC, clearance, volume of distribution, Tmax and Cmax. | From infusion of ⁸⁹Zr-Df-IAB22M2C through up to Day 6
  The data from the actual concentration and the parameters will be summarized descriptively and also presented as subject specific listings.
Evaluate the dosimetry of a single dose of ⁸⁹Zr-Df-IAB22M2C | From infusion of ⁸⁹Zr-Df-IAB22M2C through up to Day 6
  Dosimetry will be determined from the ⁸⁹Zr-Df-IAB22M2C PET/CT scans obtained during the course of this study at 1-2 hours, 6-8 hours (optional), 24 (± 4 hours), 48 (± 4 hours) hours and 92-144 hours post infusion in patients at the optimal dosing cohort. Regions of interest will be drawn at each PET/CT time point to capture target and major organ uptakes. Once all five PET/CT scans are analyzed, the biologic clearance will be evaluated from the "dynamic" sequence of the scans and the final estimated radiation dose calculated using the clearance seen in the images. The data for dosimetry also comes from Imaging Endpoints. Patterns of radiotracer uptake and estimates of semi-quantitative measurements, using typical SUV (Standardized uptake value) estimates (SUV max; SUV peak; SUV mean) will be presented. The data will be summarized descriptively and will also be presented as subject specific listings.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Honor Health and Imaging Endpoints, Scottsdale, Arizona
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Farwell MD, Gamache RF, Babazada H, Hellmann MD, Harding JJ, Korn R, Mascioni A, Le W, Wilson I, Gordon MS, Wu AM, Ulaner GA, Wolchok JD, Postow MA, Pandit-Taskar N. CD8-Targeted PET Imaging of Tumor-Infiltrating T Cells in Patients with Cancer: A Phase I First-in-Humans Study of 89Zr-Df-IAB22M2C, a Radiolabeled Anti-CD8 Minibody. J Nucl Med. 2022 May;63(5):720-726. doi: 10.2967/jnumed.121.262485. Epub 2021 Aug 19. PMID 34413145